

#### STATISTICAL REPORTING AND ANALYSIS PLAN

A randomized evaluator-blind, single-center and two-arm clinical study designed to evaluate the local tolerance and cosmetic efficacy of a topical skin care formulation in healthy female subjects with moderate to advanced photo-damaged facial skin who have undergone a 70% Glycolic Acid peel procedure

Protocol Number: 206827

Phase: NA

Property of GSK Consumer Healthcare Confidential May not be used, divulged, published or otherwise disclosed without the consent of GSK Template Version Effective: 15-Jul-2017

Page 1 of 46

## **Document History**

| Document | Version Date | Summary of Changes (New analysis or Change in planned analysis) |
|---|---|---|
| Original Analysis Plan | 12-Oct-2017 | Not applicable (N/A) |

| Ta | | f conten | | |
|---|---|---|---|---|
| | | | ory | |
| | | | nts | |
| | | • | | |
| 1 | Sumn | nary of K | ey Protocol Information | 6 |
| | 1.1 | Study D | Design | 6 |
| | 1.2 | Study C | Objectives | 6 |
| | 1.3 | Treatme | ents | 7 |
| | 1.4 | Sample | Size Calculation | 7 |
| 2 | Plann | ed Analys | ses | 7 |
| | 2.1 | Interim | Analysis | 7 |
| | 2.2 | Final A | nalyses | 8 |
| 3 | Cons | iderations | for Data Analyses and Data Handling Conventions | 8 |
| | 3.1 | Baseline | e Definition | 8 |
| | 3.2 | Subgrou | ıps/Stratifications | 8 |
| | 3.3 | Center l | Pools | 8 |
| | 3.4 | Time Po | oints and Visit Windows | 8 |
| 4 | Data . | Analysis | | 8 |
| | 4.1 | Populat | ions for Analysis | 9 |
| | | 4.1.1 | Subject Disposition | 9 |
| | | 4.1.2 | Protocol Deviations | 9 |
| | | 4.1.3 | Analysis Populations | 9 |
| | 4.2 | Subject | Demographics and Other Baseline Characteristics | 10 |
| | | 4.2.1 | Demographic Characteristics | 10 |
| | | 4.2.2 | General Medical History | 11 |
| | | 4.2.3 | Characteristics of Disease | 11 |
| | 4.3 | | ents (Study Drug/Product, Rescue Medication, other Concomitant es, Compliance) | 11 |
| | | 4.3.1 | Study Compliance and Exposure | |
| | | 4.3.2 | Prior and Concomitant Medication | |
| | 4.4 | | s of Primary and Secondary Objectives | |
| | • | 4.4.1 | Primary Objective Variable | |
| | | 4.4.2 | Secondary Objective Variables | |
| | 4.5 | | s of Safetys | |

#### Final Statistical Reporting and Analysis Plan, 12Oct2017

| | 4.5.1 Adverse Events and Serious Adverse Events | 15 |
|-----|-----------------------------------------------------------|----|
| 5 | Changes to the Protocol Defined Statistical Analysis Plan | 16 |
| 6 | Top-line Summary | 16 |
| | References | |
| | Appendix 1: Subgroups | 17 |
| | Appendix 2: Center pools in multicenter studies | |
| | Appendix 3: Major Protocol Deviations | 17 |
| Att | achment 1: List of Data Displays | |
| | Appendix 4: Templates for Tables, Figures & Listings | 19 |

Glossary

| AE | Adverse Event |
|--------|----------------------------------------------|
| BDRM | Blinded Data Review Meeting |
| CI | Confidence Interval |
| EGA | Evaluator Global Assessment |
| ITT | Intent-to-Treat |
| MedDRA | Medical Dictionary for Regulatory Activities |
| PP | Per Protocol |
| RAP | Statistical Reporting and Analysis Plan |
| TEAE | Treatment Emergent Adverse Event |
| TEWL | Transepidermal Water Loss |

The purpose of this Statistical Reporting and Analysis Plan (RAP) is to describe the planned analyses and outputs to be included in the Clinical Study Report for Protocol 206827 (version 4.0, 15-September-2017).

## 1 Summary of Key Protocol Information

The objective of this clinical study is to evaluate the local tolerance and cosmetic efficacy of a topical skin care formulation in healthy female subjects with moderate to advanced photodamaged facial skin who have undergone a 70% Glycolic Acid facial peel procedure.

### 1.1 Study Design

This is a randomized, evaluator-blind, single-center and two-arm clinical study. It is hypothesized that the test product, which is specifically designed as a moisturizing cream for dry, sensitive skin, will present a favorable local tolerance profile in this population.

### 1.2 Study Objectives

Study objectives as stated in the protocol.

| Objectives | Endpoints |
|---|---|
| Primary Objective | Primary Endpoint |
| Assessment of the local tolerance of<br>the test product in subjects who have<br>undergone a 70% Glycolic Acid<br>facial peel | Evaluator (Dermatologist) global assessment of tolerance |
| Secondary Objectives | Secondary Endpoints |
| Assessment of skin recovery (change from baseline) over a period of 14 days in subjects who have undergone a 70% Glycolic Acid facial peel | Combined (sum of) Evaluator (Dermatologist) scores for signs/symptoms of erythema, edema, desquamation and dryness Individual Evaluator (Dermatologist) scores for erythema, edema, desquamation and dryness Combined (sum of) subject self-assessment scores for redness, pain, stinging/burning, itching, tightness and dryness Individual subject self-assessment scores for redness, pain, stinging/burning, itching, tightness and dryness |

| Objectives | Endpoints |
|---|---|
| | Instrumental measurement of barrier function |
| | (Tewameter) and moisturisation |
| | (Corneometer) |
| | Subject global self-assessment |
| Assessment of skin recovery (change) | All assessments and measurements listed |
| from baseline) between treatment | above |
| groups. | |

#### 1.3 Treatments

Single test product (Physiogel Calming Relief Restoring Lipid Balm) used in combination with commercial sunscreen (Sunmax Sensitive SPF 50) and cleanser (Simple Kind to Skin Moisturising Facial Wash). Randomization was to two groups (test product, no test product) with product usage as shown in the table below:

| Randomized<br>Group | Morning | Lunchtime* | Evening |
|---|---|---|---|
| Group 1<br>(Test<br>product) | <ol> <li>Cleanser</li> <li>Test Product</li> <li>Sunscreen</li> </ol> | 1. Sunscreen | Cleanser Test Product |
| Group 2<br>(No test<br>product) | <ol> <li>Cleanser</li> <li>Sunscreen</li> </ol> | 1. Sunscreen | 1. Cleanser |

<sup>\*</sup>Lunchtime application must be at least 3 hours after previous sunscreen application

### 1.4 Sample Size Calculation

Approximately 178 healthy females within the ages of 30 and 60 years (inclusive) with Fitzpatrick Skin Classification II-IV and moderate to advanced photo-damaged skin will be screened to randomize 100 subjects to ensure approximately 80 subjects (40 subjects per group) successfully complete the study.

## 2 Planned Analyses

### 2.1 Interim Analysis

No interim analysis is planned.

### 2.2 Final Analyses

The final planned primary analyses will be performed after the completion of the following sequential steps:

- 1. All subjects have completed the study as defined in the protocol
- 2. All required database cleaning activities have been completed and database has been locked.
- 3. All criteria for unblinding the randomization codes have been met and the randomization codes have been distributed.

## 3 Considerations for Data Analyses and Data Handling Conventions

#### 3.1 Baseline Definition

The baseline for efficacy measurements and secondary assessments of local tolerance is defined as the assessments taken 60+/-15 minutes after completion of the facial peel procedure.

The primary assessment of local tolerance (EGA score, primary endpoint) is being assessed 14 days after completion of the facial peel procedure using all subjects in the safety population.

Unless otherwise stated, if baseline data is missing no derivation will be performed and will be set to missing.

#### 3.2 Subgroups/Stratifications

There was no stratification in this study.

#### 3.3 Center Pools

There was no center pool in this study.

#### 3.4 Time Points and Visit Windows

All data will be accepted for analysis. Significant numbers of deviations from the scheduled nominal visit days are not expected but in each case this occurs a protocol deviation will be recorded.

## 4 Data Analysis

Data analysis will be performed by inVentiv Health Clinical. The statistical analysis software used will be SAS version 9.4 or higher.

Prior to database closure a Blinded Data Review Meeting (BDRM) will be conducted in which various aspects of the trial will be discussed and agreed.

Except as described below, all listings will be produced for all randomized subjects.

GlaxoSmithKline Consumer Healthcare Confidential

### 4.1 Populations for Analysis

#### 4.1.1 Subject Disposition

Screen failures will be defined as subjects who do not satisfy all the inclusion/exclusion criteria. A summary will be provided of the number of subjects screened and the number of screen failures with reasons why subjects were not randomized (Table 14.1.1.1). Percentages will be based on the total number of subjects randomized.

Subject disposition will be summarized as the number and percentage of subjects (out of the number of randomized subjects) who complete the study, with the number who discontinue broken down by reason for discontinuation (Table 14.1.1.1). The table will also summarize the number and percent of subjects assigned to each analysis population (refer to section 4.1.3).

Subject disposition including the subject status (completer, Yes/No), critical demographic data (age, sex, race), the duration of treatment before discontinuation and the specific reason for discontinuation, will be listed (Listing 16.2.1.1) by treatment group.

#### 4.1.2 Protocol Deviations

Protocol deviations will be tracked by the study team throughout the conduct of the study. Data will be reviewed prior to unblinding and closure of the database to ensure all important deviations are captured and categorised.

Any deviations will be noted in the deviation log and will be evaluated to determine whether a subject exclusion from the Per Protocol population is required.

Major deviations of the protocol procedures are identified as liable to significantly influence the primary safety outcome or the key secondary efficacy outcomes (TEWL and Corneometry):

- Violation of inclusion or exclusion criteria at screening or baseline that may affect any of the above 3 assessments (Evaluator global assessment, TEWL and corneometry).
- Non-compliance with assigned treatment regimen.
- Use of prohibited treatment or medication before or during the study, which it is felt will affect any of the above 3 assessments (Evaluator global assessment, TEWL and corneometry).

The number and percentage of subjects with any major protocol deviation and with each type of major protocol deviation will be presented by treatment (Table 14.1.2) and listed (Listing 16.2.2.1). Minor protocol deviations will also be listed (Listing 16.2.2.2).

#### 4.1.3 Analysis Populations

Following analysis populations are defined.

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| Safety | All subjects with at least one application | Safety |
| | of product in the test phase (i.e. test | |

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| | <ul> <li>product for subjects in Group I or sunscreen for subjects in Group II) will be included in the Safety population.</li> <li>This population will be based on the treatment the subject actually received.</li> </ul> | |
| Intent-To-Treat | <ul> <li>All subjects who were randomized received at least one application of test product and who had at least one post-procedure post-baseline assessment will be included in the intent-to-treat (ITT) population.</li> <li>This population will be based on the treatment to which the subject was randomized.</li> </ul> | Efficacy |
| Per-Protocol | Subjects will be considered eligible for a<br>Per Protocol (PP) population if they were<br>randomized, received at least one<br>application of test product, had at least<br>one post-procedure, post-baseline<br>assessment and were compliant with both<br>test and washout products post-procedure. | Per Protocol |

The numbers of subjects included in each of the analysis populations, and the number excluded from each population broken down by the reason for exclusion will be presented (Table 14.1.2). Randomized subjects excluded from any of the analysis populations will be listed (Listing 16.2.3.1).

A PP analysis will be performed on efficacy (TEWL and Corneometry) variables only if more than 10% of the subjects in the ITT population are excluded from the PP population in any of the treatment groups.

### 4.2 Subject Demographics and Other Baseline Characteristics

Demographic and baseline characteristics summaries will be produced for the Safety, ITT and PP (if needed) populations. Dermatologist Assessment of Sensitivity and Subject Self-Assessment will be presented (Listing 16.2.6.1 and Listing 16.2.6.2).

#### 4.2.1 Demographic Characteristics

Categorical demographic variables include sex, race, Fitzpatrick and Glogau Types. These variables will be summarized by the number and percentage of subjects with each relevant characteristic in each treatment group. Age, will be summarized by the mean, standard deviation, median, minimum and maximum values in each treatment group. All demographic

information will be tabulated (Table 14.1.3.1, Table 14.1.3.2 and Table 14.1.3.3) for each population and listed (Listing 16.2.4.1) for all randomized subjects.

### 4.2.2 General Medical History

Medical history for all randomized subjects will be listed (Listing 16.2.4.2) with start date and end date or ongoing at the first application of test product.

#### 4.2.3 Characteristics of Disease

Not applicable.

# 4.3 Treatments (Study Drug/Product, Rescue Medication, other Concomitant Therapies, Compliance)

#### 4.3.1 Study Compliance and Exposure

Subjects should have at least one application of either test product or sunscreen in the test phase (from visit 3 onwards) to be included in the safety population.

Subjects identified to have no applications of product in the test phase will also be excluded from the ITT and PP population. Listings will be prepared for the BDRM only.

#### 4.3.2 Prior and Concomitant Medication

Prior medication will be defined as any medication taken prior to the first dose of study product. Concomitant medication is defined as any medication taken between the date of first dose of study product and the date of last dose of study product.

Medications missing both start and stop dates, or having a start date prior to the first dose of study product and missing the stop date, or having a stop date on or after the last dose of study product and missing start date will be counted as concomitant.

Prior and concomitant medications will be listed by subject, with preferred term, indication, dose, dose form, frequency, route, start date and start and end day (Listing 16.2.5).

### 4.4 Analysis of Primary and Secondary Objectives

#### 4.4.1 Primary Objective Variable

The primary evaluation of tolerance will be based on the safety related Evaluator (Dermatologist) global assessment. The trial will be considered a success if the majority of subjects in the test product group have a favorable ("well tolerated") Evaluator global assessment score.

The Dermatologist will assess the local tolerance of the post-procedure skin care regimen in context of the expected effects of the procedure for each subject using the scale below. To make this assessment, the Dermatologist will draw on the total set of clinical and subject self-

assessment data for each subject. The Dermatologist must be unaware of whether a subject was randomized to test product to protect the blind.

| Rating | Description |
|---|---|
| Well Tolerated | No clinically significant worsening of the expected signs/symptoms of the procedure. No new signs/symptoms manifest during product use. |
| Not Well Tolerated | Clear, clinically relevant worsening of the severity or frequency of expected signs/symptoms of the procedure and/or any occurrence of new, unexpected signs/symptoms during product use. |

#### 4.4.1.1 Statistical Hypothesis, Model, and Method of Analysis

Descriptive statistics (n, percentage, 95% confidence intervals) will be used to summarize the proportion of subjects in each product group with a favorable evaluator global assessment of tolerance and will be tabulated (Table 14.2.1.1).

Exact binomial 95% confidence intervals are calculated for the proportion well tolerated for each treatment group.

The proportions will also be compared between product groups using Chi-square test, and difference in proportion and 95% confidence interval.

#### 4.4.2 Secondary Objective Variables

Following variables are defined as secondary objective variables:

- Combined (sum of) Evaluator (Dermatologist) scores for signs/symptoms of erythema, edema, desquamation and dryness
- Individual Evaluator (Dermatologist) scores for erythema, edema, desquamation and dryness
- Combined (sum of) subject self-assessment scores for redness, pain, stinging/burning, itching, tightness and dryness
- Individual subject self-assessment scores for redness, pain, stinging/burning, itching, tightness and dryness
- Instrumental measurement of barrier function (Tewameter) and moisturisation (Corneometer)
- Subject global self-assessment

Safety measurements Evaluator (Dermatologist) and Subject assessment scores will be assessed at Baseline (60±15 minutes post-procedure), 180 minutes post-procedure, and 1, 2, 3, 7 and 14 days post-procedure.

Efficacy measurements in this study will be based on changes from baseline in TEWL and Corneometer values at each timepoint. Both measurements will be assessed pre-procedure and at Baseline (60±15 minutes post-procedure), 180 minutes post-procedure, 360 minutes post-procedure, and 1, 2, 3, 7 and 14 days post-procedure.

#### 4.4.2.1 Secondary Objective Variable 1

The sum score of the individual Evaluator Dermatologist scores will be used as safety variable. The baseline will be defined as the assessment made 60±15 minutes after the facial peel procedure, before any test product application.

#### 4.4.2.1.1 Statistical Hypothesis, Model, and Method of Analysis

Descriptive statistics will be used to summarize analyses in each product group (Table 14.2.3.1) including changes from baseline.

To visually inspect the treatment effect on dermatologist total score, a plot across time with the raw means will be produced. The plot will display a different symbol for each treatment group and presented (Figure 14.2.3.2).

Differences between product groups in the mean changes from baseline will also be explored using t-tests (different from zero) at each timepoint and summarized using 95% confidence intervals (Table 14.2.3.1).

#### 4.4.2.2 Secondary Objective Variable 2

The individual scores (erythema, edema, desquamation and dryness) of the individual Evaluator Dermatologist will be analyzed as safety variable.

#### 4.4.2.2.1 Statistical Hypothesis, Model, and Method of Analysis

The individual scores of the individual Evaluator Dermatologist will be defined as the assessment made 60±15 minutes after the facial peel procedure, before any test product application and presented separately for each individual score (Table 14.2.3.4, Table 14.2.3.5, Table 14.2.3.6 and Table 14.2.3.7) including changes from baseline.

Summary stats and frequency counts will be presented (Table 14.2.3.2) for all individual scores and to be used if sufficient data is not available for formal analyses for individual score.

Differences between product groups in the mean changes from baseline will also be explored using t-tests (different from zero) at each timepoint and summarized using 95% confidence intervals (Table 14.2.3.4, Table 14.2.3.5, Table 14.2.3.6 and Table 14.2.3.7) separately for each of those individual scores.

#### 4.4.2.3 Secondary Objective Variable 3

The sum score subject self-assessment scores will be analyzed as safety variable. The baseline will be defined as the assessment made 60±15 minutes after the facial peel procedure, before any test product application.

#### 4.4.2.3.1 Statistical Hypothesis, Model, and Method of Analysis

Descriptive statistics will be used to summarize analyses in each product group (Table 14.2.2.1) including changes from baseline.

To visually inspect the treatment effect on subject self-assessment total score, a plot across time with the raw means will be produced. The plot will display a different symbol for each treatment group and presented (Figure 14.2.2.2).

Differences between product groups in the mean changes from baseline will also be explored using t-tests (different from zero) at each timepoint and summarized using 95% confidence intervals (Table 14.2.2.1).

#### 4.4.2.4 Secondary Objective Variable 4

The individual scores (redness, pain, stinging/burning, itching, tightness and dryness) of the subject self-assessment will be analyzed as safety variable.

#### 4.4.2.4.1 Statistical Hypothesis, Model, and Method of Analysis

The individual scores of the subject self-assessment will be defined as the assessment made 60±15 minutes after the facial peel procedure, before any test product application and presented separately for each individual score (Table 14.2.2.4, Table 14.2.2.5, Table 14.2.2.6, Table 14.2.2.7, Table 14.2.2.8 and Table 14.2.2.9) including changes from baseline.

Summary stats and frequency counts will be presented (Table 14.2.2.2) for all individual scores and to be used if sufficient data is not available for formal analyses for individual score.

Differences between product groups in the mean changes from baseline will also be explored using t-tests (different from zero) at each timepoint and summarized using 95% confidence intervals (Table 14.2.3.4, Table 14.2.3.5, Table 14.2.3.6 and Table 14.2.3.7) separately for each of those individual scores.

#### 4.4.2.5 Secondary Objective Variable 5

Instrumental measurement of barrier function (Tewameter) and moisturisation (Corneometer) are efficacy related variables.

A PP analysis will be performed on those variables (Table 14.2.4.2 and Table 14.2.5.2) only if more than 10% of the subjects in the ITT population are excluded from the PP population in any of the treatment groups.

#### 4.4.2.5.1 Statistical Hypothesis, Model, and Method of Analysis

Changes from baseline in instrumental endpoints (TEWL and corneometry) will be tabulated by product group and timepoint and summarized descriptively and presented (Table 14.2.4.1 and Table 14.2.5.1).

Differences between product groups in the mean changes from baseline will also be explored using t-tests (different from zero) at each timepoint and summarized using 95% confidence intervals (Table 14.2.4.1 and Table 14.2.5.1) separately for each of those two variables.

#### 4.4.2.6 Secondary Objective Variable 6

Subject global assessment of satisfaction evaluated at the last post-procedure follow-up visit (Day 22 – 14 days post-procedure) will be analyzed as efficacy related variable (Table 14.2.6.1).

#### 4.4.2.6.1 Statistical Hypothesis, Model, and Method of Analysis

Subject global assessment of satisfaction will be summarized by product group and tabulated for each rating descriptively using N and percentage of subjects. The ratings of "Total Satisfied" and "Very Satisfied" will also be combined and summarized descriptively (N, percent of subjects) by product group (Table 14.2.6.1).

Exact binomial 95% confidence intervals are calculated for the proportion of total satisfied and very satisfied (Table 14.2.6.1).

The difference between product groups in the proportion of "Total Satisfied" and "Very Satisfied" subjects will also be presented with a 95% confidence interval for the difference and evaluated for a treatment difference via Chi-square test (Table 14.2.6.1).

#### 4.5 Analysis of Safety

#### 4.5.1 Adverse Events and Serious Adverse Events

Treatment emergent adverse events (TEAEs) are defined as events that start on or after the first product application in the test phase.

Adverse events (AEs) will be coded according to the current version of the Medical Dictionary for Regulatory Activities (MedDRA). Frequencies and percentages will be presented by product group and overall, for each system organ class, and for each preferred term.

All TEAEs will be summarized by the number and percentage of subjects having any AE, an adverse event in each system organ class, and each individual AE (Table 14.3.1.1). All TEAEs will also be tabulated by severity (Table 14.3.1.3). TEAEs suspected of a relationship to study medication and those causing study discontinuation will be presented in a similar manner (Table 14.3.1.2 and Listing 14.3.2.6).

Additionally, all adverse events will be listed (Listing 16.2.7.1 and Listing 16.2.7.2).

Deaths occurring during treatment (if any) will be listed by treatment, including the date and study day of death, and the principal cause of death (Listing 14.3.2.1). Non-fatal serious AEs

and AEs causing study treatment discontinuation will be listed (Listing 14.3.2.2 and Listing 14.3.2.3).

### 5 Changes to the Protocol Defined Statistical Analysis Plan

There are no changes to the protocol-planned statistical analyses. However, if there is no sufficient data available for formal analysis, summary stats and frequency counts will be presented.

## **6** Top-line Summary

For the top-line report selected outputs will be produced as documented in the attached worksheet excel file

#### 7 References

None

Appendix 1: Subgroups

Not Applicable

Appendix 2: Center pools in multicenter studies

Not Applicable

## **Appendix 3: Major Protocol Deviations**

Protocol deviations will be tracked by the study team throughout the conduct of the study. All violations will be reviewed prior to study unblinding and closure of the database. Details will be given in the populations' definitions document.



## Attachment 1: List of Data Displays





### Appendix 4: Templates for Tables, Figures & Listings

This is a guideline which will give the guidance of treatment labels that will be used for the table header and in the figures, listings and in the footnotes.

The treatment labels for the column heading will be as follow:

- Physiogel Calming Relief Restoring Lipid Balm
- No Test Product

If there are no data to display generate a null table or listing.



#### Final Statistical Reporting and Analysis Plan, 12Oct2017

Protocol No. 206827 Page x of y
Program Run Date:xxxx

# Table 14.1.1.1 Subject Disposition by Treatment Group All Screened Subjects

All Screened Subjects (N=xxx)

| | Physiogel Calming Relief<br>Restoring Lipid Balm | No Test Product | Overall |
|---|---|---|---|
| | N (%) | N (%) | N (%) |
| | 2. (0) | 1. (0) | 4 (0) |
| TOTAL SUBJECTS SCREENED | | | xxx |
| SUBJECTS NOT RANDOMIZED | | | xxx |
| DID NOT MEET STUDY CRITERIA | | | xxx (xx.x) |
| ADVERSE EVENT | | | Xxx (xx.x) |
| LOST TO FOLLOW UP | | | xxx (xx.x) |
| PROTOCOL VIOLATION | | | Xxx (xx.x) |
| WITHDRAWAL OF CONSENT | | | Xxx (xx.x) |
| OTHER | | | Xxx (xx.x) |
| SUBJECTS RANDOMIZED | xxx | xxx | xxx |
| COMPLETED STUDY | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| DID NOT COMPLETE STUDY | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| DID NOT MEET STUDY CRITERIA | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| ADVERSE EVENT | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| LOST TO FOLLOW-UP | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| PROTOCOL VIOLATION | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| WITHDRAWAL OF CONSENT | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| OTHER | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| SAFETY POPULATION | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| ITT POPULATION | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| PP POPULATION | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |

Program file name xxxxxxxxxxxxxxxxx

Programming note: For categories under 'Subjects Not Randomized' percentages will be calculated using the number of 'All Screened Subjects' as the denominator. Percentages under the 'Subjects Randomized' categories will be computed using number of subjects randomized as the denominator.



#### Final Statistical Reporting and Analysis Plan, 12Oct2017

Protocol No. 206827

Page x of y
Program Run Date:xxxx

Table 14.1.2

Analysis of Population
All Randomized Subjects

Randomized Population (N=xxx)

| | Physiogel Calming Relief | No Test Product | 0veral1 |
|---|---|---|---|
| | Restoring Lipid Balm N (%) | N (%) | N (%) |
| UBJECTS EXCLUDED FROM SAFETY POPULATION | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| REASON 1 | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| ••• | | | |
| UBJECTS EXCLUDED FROM ITT POPULATION | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| REASON 1 | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| UBJECTS WITH AT LEAST ONE DATA POINT EXCLUDED ROM PP ANALYSIS | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| UBJECTS COMPLETELY EXCLUDED FROM PP POPULATION | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| ROTOCOL DEVIAIONS LEADING TO EXCLUSION FROM PP | | | |
| CCLUDING ALL | | | |
| DEVIATION 1 | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| ••• | | | |
| KCLUDING WEEK X | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| DEVIATION X | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |



#### Final Statistical Reporting and Analysis Plan, 12Oct2017

Program Run Date:xxxx

Table 14.1.3.1 Demographics Safety Population

ITT Population (N=xxx)

| | Physiogel Calming Relief | | |
|---|---|---|---|
| | Restoring Lipid Balm | No Test Product | Overall |
| | (N=xx) | (N=xx) | (N=xxx) |
| SEX n (%) | | | |
| FEMALE | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| RACE n (%) | | | |
| AMERICAN INDIAN OR ALASKA NATIVE | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ASIAN | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| BLACK OR AFRICAN AMERICAN | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| NATIVE HAWAIIAN OR OTHER PACIFIC ISLANDER | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| WHITE | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| MULTIPLE | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| AGE (YEARS) | | | |
| N | xx | xx | xx |
| MEAN | xx.x | xx.x | xx.x |
| SD | xx.xx | xx.xx | xx.xx |
| MEDIAN | xx.x | xx.x | xx.x |
| MINIMUM | xx | xx | xx |
| MUMIXAM | xx | xx | xx |
| FITZPATRICK PHOTOTYPE n (%) | | | |
| I | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| II | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| III | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| GLOGAU PHOTOTYPE n (%) | | | |
| I | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| II | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| III | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| IV | xx (xx.x) | xx (xx.x) | xx (xx.x) |



#### Final Statistical Reporting and Analysis Plan, 12Oct2017

Program Run Date:xxxx

# Table 14.2.1.1 Summary of Evaluator Global Assessment Score Safety Population

Safety Population (N=xx)

| | Physiogel Calming Relief<br>Restoring Lipid Balm | No Test Product |
|---|---|---|
| | (N=xx) | (N=xx) |
| n | xx | xx |
| Missing | XX (XX%) | XX (XX%) |
| Product Regimen was Well Tolerated | XX (XX%) | XX (XX%) |
| Product Regimen was Not Well Tolerated | XX (XX%) | XX (XX%) |
| 95% Confidence Interval for Proportion Well Tolerated | (XX.X%, XX.X%) | (XX.X%, XX.X%) |
| Difference in Proportions Well Tolerated (95% Confidence Interval) | xx% (xx.x - | - xx.x) |
| Chi-Square P-Value | x.xx | K |



#### Final Statistical Reporting and Analysis Plan, 12Oct2017

Program Run Date:xxxx

 $\begin{tabular}{ll} Table 14.2.3.1 \\ Summary of Dermatologist Assessments - Total Score \end{tabular}$ 

| Safety | 7 Popul | ation | (N=xx) | ١ |
|--------|---------|-------|--------|---|
|--------|---------|-------|--------|---|

| Timepoint | | Physiogel Calming Relief<br>Restoring Lipid Balm | No Test Product |
|---|---|---|---|
| - | | (N=xx) | (N=xx) |
| Pre-Procedure Assessment | n | xx | XX |
| | Missing | XX | XX |
| | Mean | x.xx | x.xx |
| | SD | x.xxx | x.xxx |
| | 95%CI | x.xx, x.xx | x.xx, x.xx |
| Baseline* | n | XX | xx |
| | Missing | XX | xx |
| | Mean | x.xx | x.xx |
| | SD | x.xxx | x.xxx |
| | 95%CI | x.xx, x.xx | x.xx, x.xx |
| 180 Minutes Post-Procedure | n | XX | xx |
| | Missing | XX | xx |
| | Mean | x.xx | x.xx |
| | SD | x.xxx | x.xxx |
| | 95%CI | x.xx, x.xx | x.xx, x.xx |
| Change from Baseline at 180 | n | XX | xx |
| Minutes | Missing | XX | xx |
| | Mean | x.xx | x.xx |
| | SD | x.xxx | x.xxx |
| | 95%CI | x.xx, x.xx | x.xx, x.xx |
| | P-Value* | x.xxx | x.xxx |
| Difference between Groups at 180<br>Minutes | Difference<br>(95%CI) | X.XX (X.XX, X | .XX) |
| | P-Value <sup>\$</sup> | x.xxx | |



#### Final Statistical Reporting and Analysis Plan, 12Oct2017

- <sup>8</sup> Total score=sum of Erythema, Dryness, Desquamation/Peeling and Edema individual scores.
- \* P-value from t-test compared to zero.
- \$ P-value from t-test(pooled variances).
- \* Baseline score is assessed 60 minutes post-procedure and prior to any test product application.

Program file name xxxxxxxxxxxxxxxxxx

#### Programmer Note:

Change the title, footnote and time points to match protocol for other tables with same layout. For individual scores no footnote about total scores.



Final Statistical Reporting and Analysis Plan, 12Oct2017

Program Run Date:xxxx

Figure 14.2.3.2

Dermatologist Assessment Scores - Total Score
Safety Population

PPD

Safety Population

Program file name xxxxxxxxxxxxxxxxxx

Programmers Note: Figure to be created for Safety population.

Change the title, footnote and time points to match protocol and adapt reference table. Adapt also correct treatment description.



#### Final Statistical Reporting and Analysis Plan, 12Oct2017

Program Run Date:xxxx

Table 14.2.3.3 Summary of Dermatologist Assessments - Individual Assessments Safety Population

Safety Population (N=xx)

| | Pl | Physiogel Calming Relief Restoring Lipid Balm (N=xx) | | | | | | | No Test Product<br>(N=xx) | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Missing | None | Mild | Moderate | Severe | Total | Missing | None | Mild | Moderate | Severe | Total |
| Erythema | | | | | | | | | | | | |
| Pre-<br>procedure | X (xx%) | X(xx%) | X (xx%) | X(xx%) | X (xx%) | Х | X(xx%) | X (xx%) | X(xx%) | X (xx8) | X(xx%) | х |
| | X (xx%) | X(xx%) | X (xx%) | X(xx%) | X (xx%) | x | X(xx%) | X(xx <sup>8</sup> ) | X(xx%) | X (xx%) | X (xx%) | х |
| Baseline* | | | | | | | | | | | | |
| Score | | | | | | | | | | | | |
| 180 Min | X(xx%) | X(xx%) | X(xx%) | X(xx%) | X(xx%) | X | X(xx%) | X (xx%) | X(xx%) | X(xx%) | X(xx%) | x |
| 1 Day | X (xx%) | X(xx%) | X(xx%) | X(xx%) | X(xx%) | Х | X(xx%) | X (xx%) | X(xx%) | X(xx%) | X(xx%) | x |
| 2 Days | X(xx%) | X(xx%) | X(xx%) | X(xx%) | X(xx%) | X | X(xx%) | X (xx%) | X(xx%) | X(xx%) | X(xx%) | x |
| 3 Days | X(xx%) | X(xx8) | (xx%) | X(xx%) | X (xx8) | X | X (xx%) | X(xx%) | X(xx%) | X (xx%) | X (xx%) | х |
| 7 Days | X (xx%) | X(xx8) | X<br>(xx%) | X (xx8) | X (xx8) | X | X (xx8) | X (xx%) | X(xx%) | X (xx%) | X (xx%) | х |
| 14 Days | X (xx%) | X<br>(xx%) | X<br>(xx%) | X(xx%) | X (xx%) | х | X(xx8) | X (xx <sup>8</sup> ) | X(xx8) | X (xx%) | X (xx%) | х |
| <other td="" war<=""><td>iables&gt;</td><td></td><td></td><td></td><td></td><td></td><td></td><td></td><td></td><td></td><td></td><td></td></other> | iables> | | | | | | | | | | | |

<sup>\*</sup> Baseline score is assessed 60 minutes post-procedure and prior to any test product application.

Percentages based on total number of subjects per product group.

Program file name xxxxxxxxxxxxxxxxxx

Programmer's note: Same format for other table (change assessments to match protocol). Repeat for other individual variables with same time points within table



#### Final Statistical Reporting and Analysis Plan, 12Oct2017

Program Run Date:xxxx

Table 14.2.6.1

Summary of Subjects Global Assessment of Satisfaction
Intent-to-Treat Population

#### ITT Population(N=xx)

| | Physiogel Calming Relief<br>Restoring Lipid Balm | No Test Product |
|---|---|---|
| | (N=xx) | (N=xx) |
| n | xx | xx |
| Missing | XX (XX%) | XX (XX%) |
| Very Satisfied | XX (XX%) | XX (XX%) |
| Satisfied | XX (XX%) | XX (XX%) |
| - Total Satisfied and Very Satisfied | XX (XX%) | XX (XX%) |
| 95% Confidence Interval (Total Satisfied and Very Satisfied) | XX.X%, XX.X% | xx.x%, xx.x% |
| Difference in Proportions Total Satisfied | xx% (xx.x - | - XX.X) |
| and Very Satisfied (95% Confidence Interval) | | |
| Chi-Square P-Value | x.xxx | ( |
| Poorly Satisfied | XX (XX%) X | X (XX%) |
| Not at all Satisfied | XX (XX%) | X (XX%) |

Percentages based on total number of subjects per product group.

Exact binomial 95% confidence intervals are calculated for the proportion of total satisfied and very satisfied.



#### Final Statistical Reporting and Analysis Plan, 12Oct2017


Page x of y
Program Run Date:xxxx

# Table 14.3.1.1 Treatment Emergent Adverse Events Safety Population

Safety Population (N=xx)

| | Physiogel Calming Relief<br>Restoring Lipid Balm<br>(N=XX) | No Test Product (N=XX) | Overall (N=XXX) |
|---|---|---|---|
| | n (%) nAE | n (%) nAE | n (%) nAE |
| NUMBER OF SUBJECTS WITH AT LEAST ONE AE NUMBER OF SUBJECTS WITH NO AE | xx ( xx.x) xx | xx ( xx.x) xx | xx ( xx.x) xx |
| | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) |
| SOC1 | xx ( xx.x) xx | xx ( xx.x) xx | xx ( xx.x) xx |
| PT1 | xx ( xx.x) xx | xx ( xx.x) xx | xx ( xx.x) xx |
| SOC2 | xx ( xx.x) xx | xx ( xx.x) xx | xx ( xx.x) xx |
| PT1 | xx ( xx.x) xx | xx ( xx.x) xx | xx ( xx.x) xx |

Programmer's note: Same format for other table

n (%) = Number (percent) of subjects nAE = Number of adverse events. SOC: System of Organ Class Program file name xxxxxxxxxxxxxxxxxxx



#### Final Statistical Reporting and Analysis Plan, 12Oct2017


Page x of y
Program Run Date:xxxx

# ${\small \mbox{Table 14.3.1.3}}$ Summary of Treatment Emergent Adverse Event by Severity ${\small \mbox{Safety Population}}$

| Safety Population (N=xx) | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| System of Organ Class (SOC) Preferred Term (PT) | Physio | gel Cal | ming Relie | f Resto | ring Lipid Balm | n | No Te | st Prod | luct | | | |
| | | | (N= | XX) | | | | (N=XX) | | | | |
| | Mild | | Moderate | | Severe | | Mild | | Moder | ate | Severe | |
| | n (%) | nAE | n (%) | nAE | n (%) | nAE | n (%) | nAE | n (%) | nAE | n (%) | nAE |
| NUMBER OF SUBJECTS WITH AT LEAST ONE AE | xx (xx.x) | xx | xx<br>(xx.x) | xx | xx (xx.x) | xx | xx (xx.x) | xx | **<br>(**.*) | xx | xx (xx.x) | xx |
| SOC1 | xx (xx.x) | xx | xx<br>(xx.x) | xx | xx (xx.x) | xx | xx (xx.x) | xx | xx<br>(xx.x) | xx | xx (xx.x) | xx |
| PT1 | xx (xx.x) | xx | xx<br>(xx.x) | xx | xx (xx.x) | xx | xx (xx.x) | xx | xx<br>(xx.x) | xx | xx (xx.x) | xx |
| PT2 | xx (xx.x) | xx | xx<br>(xx.x) | xx | xx (xx.x) | xx | xx (xx.x) | xx | xx<br>(xx.x) | xx | xx (xx.x) | xx |
| PT3 | xx (xx.x) | xx | xx<br>(xx.x) | xx | xx (xx.x) | xx | xx (xx.x) | xx | xx<br>(xx.x) | xx | xx (xx.x) | xx |
| SOC2 | xx (xx.x) | xx | xx<br>(xx.x) | xx | xx (xx.x) | xx | xx (xx.x) | xx | xx<br>(xx.x) | xx | xx (xx.x) | xx |
| PT1 | xx (xx.x) | xx | xx<br>(xx.x) | xx | xx (xx.x) | xx | xx (xx.x) | xx | xx<br>(xx.x) | xx | xx (xx.x) | xx |
| PT2 | xx (xx.x) | xx | xx<br>(xx.x) | xx | xx (xx.x) | xx | xx (xx.x) | xx | xx<br>(xx.x) | xx | xx (xx.x) | xx |
| PT3 | xx (xx.x) | xx | xx<br>(xx.x) | xx | xx (xx.x) | xx | xx (xx.x) | xx | xx<br>(xx.x) | xx | xx (xx.x) | xx |

n (%) = Number (percent) of subjects nAE = Number of adverse events.

Programmer's note: Same format for other table



Program Run Date:xxxx

Listing 16.1.7.1
Randomization Details
All Randomized Subjects

| Subject Number | Age/Sex/Race [1] | Randomization Number | Randomized Treatment | Randomization Date |
|---|---|---|---|---|
| PPD | | PPD | | |

<sup>[1]</sup> Age in years; Sex: F = Female, M = Male; Race: A = Asian, B = Black or African American, I = American Indian or Alaska Native, H = Native Hawaiian or Other Pacific Islander, W = White, M = Multiple.



#### Final Statistical Reporting and Analysis Plan, 12Oct2017


Page x of y
Program Run Date:xxxx

Listing 16.2.1.1
Subject Disposition
All Randomized Subjects

#### Treatment Group: XXXXX

| | | | Treatment | Date of | Duration of | | | |
|---|---|---|---|---|---|---|---|---|
| | Sex/Age/ | Screening | Start Date | Completion or | Treatment | Completed | | |
| Subject | Race [1] | Date | and Time | Withdrawal | (Days) | (Yes/No) | Primary Reason for Withdrawal | Further Details [2] |

## PPD

[1] Age in years; Sex: F = Female, M = Male; Race: A = Asian, B = Black or African American, I = American Indian or Alaska Native, H = Native Hawaiian or Other Pacific Islander, W = White, M = Multiple.

[2] Further details of reasons for withdrawal.



#### Final Statistical Reporting and Analysis Plan, 12Oct2017


Page x of y
Program Run Date:xxxx

Listing 16.2.1.2 Subject Disposition Non-Randomized Subjects

Sex/Age/ Screening
Subject Race [1] Date Reason for Screen Failure Further Details [2]
PPD

<sup>[1]</sup> Age in years; Sex: F = Female, M = Male; Race: A = Asian, B = Black or African American, I = American Indian or Alaska Native, H = Native Hawaiian or Other Pacific Islander, W = White, M = Multiple.

<sup>[2]</sup> Further details of reasons for screen failure.



Program Run Date:xxxx

Listing 16.2.2.1

Major Protocol Deviations
All Randomized Subjects

Treatment Group: XXXXXX

| Subject | Sex/Age/ Race [1] | Week(s)<br>Excluded from<br>PP Population | Deviation<br>Reason |
|---|---|---|---|
| PPD | | All | Inclusion criteria |
| | | From Week 4 | Inclusion criteria |
| | | Week 8 | No post-baseline efficacy data available |
| | | xx | Exclusion criteria |
| | | xx | Additional uses of washout product prior to randomisation |

[1] Age in years; Sex: F = Female, M = Male; Race: A = Asian, B = Black or African American, I = American Indian or Alaska Native, H = Native Hawaiian or Other Pacific Islander, W = White, M = Multiple.

Programming Note: Listing 16.2.2.1 lists only those identified in population definition document.



#### Final Statistical Reporting and Analysis Plan, 12Oct2017

Program Run Date:xxxx

Listing 16.2.2.2

Minor Protocol Deviations

Randomized Population

<sup>[1]</sup> Age in years; Sex: F = Female, M = Male; Race: A = Asian, B = Black or African American, I = American Indian or Alaska Native, H = Native Hawaiian or Other Pacific Islander, W = White, M = Multiple.



#### Final Statistical Reporting and Analysis Plan, 12Oct2017


Page x of y
Program Run Date:xxxx

# Listing 16.2.3.1 Exclusions from Analysis Populations All Randomized Subjects

Treatment Group: XXXX

| | Sex/Age/ Race [1] | Randomized | Safety | ITT | Per Protocol |
|---|---|---|---|---|---|
| Subject | | (Yes/No) | (Yes/No) | (Yes/No) | (Yes/No) |
| PPD | | | | | |
| | | Yes | YES | YES | No |

<sup>[1]</sup> Age in years; Sex: F = Female, M = Male; Race: A = Asian, B = Black or African American, I = American Indian or Alaska Native, H = Native Hawaiian or Other Pacific Islander, W = White, M = Multiple.



#### Final Statistical Reporting and Analysis Plan, 12Oct2017


Page x of y
Program Run Date:xxxx

# Listing 16.2.4.1 Demographic Characteristics All Randomized Subjects

Treatment Group: XXXXX

| Subject | Sex | Race | Age (years) | Fitzpatrick Skin Type | Glogau Photoaging Type |
|---|---|---|---|---|---|
| PPD | | | | | |



#### Final Statistical Reporting and Analysis Plan, 12Oct2017


Page x of y
Program Run Date:xxxx

Listing 16.2.4.2

Medical History

All Randomized Subjects

| Treatment Group: | XXXXX |
|------------------|-------|
|------------------|-------|

| Subject | Sex/Age/<br>Race [1] | Any Medical<br>History?<br>(Yes/No) | Medical Condition | Medical Condition Start Date | | Ongoing? (Yes/No) End Date |
|---|---|---|---|---|---|---|
| _Subject<br>PPD | | | xxxxxxxxxx | | No | |

[1] Age in years; Sex: F = Female, M = Male; Race: A = Asian, B = Black or African American, I = American Indian or Alaska Native, H = Native Hawaiian or Other Pacific Islander, W = White, M = Multiple.

Page x of y



#### Final Statistical Reporting and Analysis Plan, 12Oct2017


Page x of y
Program Run Date:xxxx

# Listing 16.2.5 Prior and Concomitant Medication All Randomized Subjects

| Treatment 0 | Treatment Group: XXXXX | | | | | | |
|---|---|---|---|---|---|---|---|
| Subject<br>Number | Age/Sex/Race[ | 1] Concomitant?<br>[2] | Treatment | Reason for<br>Treatment | Frequency | Start Date<br>(Study Day<br>[3]) | End Date/Ongoing |
| PPD | | No | xxxxx | xxxxx | xx | Jul2017 (xx) | Ongoing |
| | | Yes | xxxxx | xxxxx | xx | Jun2017 (xx) | ddmmmyyy |

<sup>[1]</sup> Age in years; Sex: F = Female, M = Male; Race: A = Asian, B = Black or African American, I = American Indian or Alaska Native, H = Native Hawaiian or Other Pacific Islander, W = White, M = Multiple.

<sup>[2]</sup> Concomitant medication defined as <definition from the RAP>.

<sup>[3]</sup> Study day relative to the date of randomization.



#### Final Statistical Reporting and Analysis Plan, 12Oct2017


Page x of y
Program Run Date:xxxx

Listing 16.2.6.1 Subject Self-Assessment All Randomized Subjects

Treatment Group: XXXXXX
Sex/Age/

| Subject | Sex/Age/<br>Race [1] | Visit | Visit<br>Date | Variable | Observed<br>Value | Change from Baselir |
|---|---|---|---|---|---|---|
| PD | | | | | | |

[1] Age in years; Sex: F = Female, M = Male; Race: A = Asian, B = Black or African American, I = American Indian or Alaska Native, H = Native Hawaiian or Other Pacific Islander, W = White, M = Multiple.

O=None; 1=Mild; 2=Moderate; 3=Severe

Total Score = Sum of all individual scores.

Program file name xxxxxxxxxxxxxxxxx

Programmer Note: please include post baseline time points in chronological order and use same list of variables



#### Final Statistical Reporting and Analysis Plan, 12Oct2017


Page x of y
Program Run Date:xxxx

# Listing 16.2.6.2 Dermatologist Assessment All Randomized Subjects

| Assessment | | | |
|---|---|---|---|
| Variable | Score | Decode | Description |
| Erythema | 0 | None | No evidence of erythema present |
| | 1 | Mild | Slight red coloration |
| | 2 | Moderate | Definite redness |
| | 3 | Severe | Marked erythema, bright red to dusky dark red in color |
| _ | | | |
| Dryness | 0 | None | No dryness |
| | 1 | Mild | Barely perceptible, fine scales or flakes present to limited areas of the test site |
| | 2 | Moderate | Fine scales or flakes generalized to all areas of the test site |
| | 3 | Severe | Scaling and peeling of skin over all areas of the test site |
| <other></other> | | | |

Program file name xxxxxxxxxxxxxxxxx

Programmer Note: please add |other| assessment variables according to CRF Programmer Note: this is page 1 of the shell



#### Final Statistical Reporting and Analysis Plan, 12Oct2017


Treatment Group: XXXXXX

Sex/Age/

Page x of y Program Run Date:xxxx

#### Listing 16.2.6.2 Dermatologist Assessment All Randomized Subjects

Observed

PPD

Subject Race [1] Visit Date Variable Value Change from Baseline

Visit

[1] Age in years; Sex: F = Female, M = Male; Race: A = Asian, B = Black or African American, I = American Indian or Alaska Native, H = Native Hawaiian or Other Pacific Islander, W = White, M = Multiple. Total Score = Sum of all individual scores.

Program file name xxxxxxxxxxxxxxxxx

Programmer Note: this is page 2 of the shell

Programmer Note: please include post baseline time points in chronological order and use same list of variables

Programmer Note: change from baseline for all variables



#### Final Statistical Reporting and Analysis Plan, 12Oct2017

Visit

Program Run Date:xxxx

# Listing 16.2.6.3 Transepidermal Water Loss (TEWL) All Randomized Subjects

Treatment Group: XXXXXX

Sex/Age/ Visit

Variable Observed (g/m2/hr) Value Change from Baseline

#### Subject PPD

[1] Age in years; Sex: F = Female, M = Male; Race: A = Asian, B = Black or African American, I = American Indian or Alaska Native, H = Native Hawaiian or Other Pacific Islander, W = White, M = Multiple.

TEWL: Transepidermal Water Loss

Race [1]

Program file name xxxxxxxxxxxxxxxxx

Programmer Note: please include post baseline time points in chronological order and use same list of variables Programmer Note: change from baseline only to be calculated for the mean score



#### Final Statistical Reporting and Analysis Plan, 12Oct2017


Page x of y
Program Run Date:xxxx

# Listing 16.2.6.4 Corneometry All Randomized Subjects

Treatment Group: XXXXXX

| Sex/Age/ | | Visit | | Observed | Change from |
|------------------|-------|-------|----------|----------|-------------|
| Subject Race [1] | Visit | Date | Variable | Value | Baseline |

### PPD

[1] Age in years; Sex: F = Female, M = Male; Race: A = Asian, B = Black or African American, I = American Indian or Alaska Native, H = Native Hawaiian or Other Pacific Islander, W = White, M = Multiple.

Program file name xxxxxxxxxxxxxxxxx

Programmer Note: please include post baseline time points in chronological order and use same list of variables Programmer Note: change from baseline only to be calculated for the mean score



#### Final Statistical Reporting and Analysis Plan, 12Oct2017

Program Run Date:xxxx

Listing 16.2.7.1

Adverse Events

All Randomized Subjects

| Treatment G | Treatment Group: XXXXXX | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject<br>Number | Age/<br>Sex/<br>Race[1] | Adverse Event (Preferred Term) [System of Organ Class] | Start Date<br>(Study<br>Day)[2] | Start<br>Time | End Date | End<br>Time | Frequency/<br>Intensity[3] | Related<br>to Study<br>Product? | Action<br>Taken re<br>Study<br>Product | Outcome | Seri<br>ous? | With-<br>drew?<br>[4] |
| -PPD | | Headache | 31MAR2017(3) | 9:00 | 31MAR2017 | 11:00 | INT/Mild | No | | | No | No |

Program file name xxxxxxxxxxxxxxxxxx

Programmer's note: Same format for other listings

<sup>[1]</sup> Age in years; Sex: F = Female, M = Male; Race: A = Asian, B = Black or African American, I = American Indian or Alaska Native, H = Native Hawaiian or Other Pacific Islander, W = White, M = Multiple.

<sup>[2]</sup> Study day is the day relative to start of treatment, day 1 being the day of first treatment.

<sup>[3]</sup> INT = Intermittent and SGLE = Single.

<sup>[4]</sup> Did subject withdraw from study as a result of this adverse event?



#### Final Statistical Reporting and Analysis Plan, 12Oct2017


Page x of y
Program Run Date:xxxx

# Listing 16.2.7.2 Adverse Events Non-Randomized Subjects

| Subject<br>Number | Age/<br>Sex/<br>Race[1] | Adverse Event<br>(Preferred<br>Term)<br>[System of<br>Organ Class] | Start Date | Start<br>Time | End Date | End<br>Time | Frequency/<br>Intensity[2] | Related<br>to Study<br>Product? | Action<br>Taken re<br>Study<br>Product | Outcome | Seri<br>ous? | With-<br>drew?<br>[3] |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| PPD | | Headache | 31MAR2017 | 9:00 | 31MAR2017 | 11:00 | INT/Mild | No | | | No | No |

<sup>[1]</sup> Age in years; Sex: F = Female, M = Male; Race: A = Asian, B = Black or African American, I = American Indian or Alaska Native, H = Native Hawaiian or Other Pacific Islander, W = White, M = Multiple.

<sup>[2]</sup> INT = Intermittent and SGLE = Single.

<sup>[3]</sup> Did subject withdraw from study as a result of this adverse event?